CLINICAL TRIAL: NCT02939261
Title: Guelph Family Health Study: Full Study
Acronym: GFHS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Jess Haines, Associate Professor/GFHS Associate Director, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14AP009
Record Dates: First submitted 2016-10-13; First posted 2016-10-20 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Families randomized to control will receive monthly emails containing publicly available handouts on general child health.
  Interventions: Behavioral: Control
- Intervention - 4 Home Visits (Experimental): Families randomized to the intervention will receive: a) 4 home visits from a health educator, b) weekly e-mails, and c) monthly mailed behavioural supports.
  Interventions: Behavioral: Intervention - 4 Home Visits

INTERVENTIONS:
Behavioral: Intervention - 4 Home Visits — 4 home visits from a health educator, weekly e-mails, and monthly mailed behavioural supports.
  Arms: Intervention - 4 Home Visits
Behavioral: Control — monthly emails with general health information
  Arms: Control

SUMMARY:
The overall objective of this research is to test, among families with children age 2-5 years, the immediate and longer-term impacts of a home-based intervention to improve household routines associated with reduced obesity risk. The investigators primary hypothesis is that, compared to control, children in the intervention group will have lower BMI following the 6-month intervention period and 18-month follow-up period. The secondary outcomes are change in children's % body fat, waist circumference and obesity-related behaviours: sleep, activity, sedentary behaviour, family meals, and dietary intake. Although child outcomes are the focus of this evaluation, changing household routines may also improve parent behaviour; thus, the investigators will assess change in parent behaviours and weight outcomes. This study will also assess the cost-effectiveness of the intervention from a societal perspective.

DETAILED DESCRIPTION:
The overall objective of this research is to test, among families with children age 2-5 years, the immediate and longer-term impacts of a home-based intervention to improve household routines associated with reduced obesity risk. The primary hypothesis is that, compared to control, children in the intervention group will have lower BMI following the 6-month intervention period and 18-month follow-up period. The secondary outcomes are change in children's % body fat, waist circumference and obesity-related behaviours: sleep, activity, sedentary behaviour, family meals, and dietary intake. Although child outcomes are the focus of this evaluation, changing household routines may also improve parent behaviour; thus, the investigators will assess change in parent behaviours and weight outcomes. This study also assess the cost-effectiveness of the intervention from a societal perspective.

The investigators will randomly allocate 356 socio-economically diverse Ontario families to receive either: 1) 4 motivational coaching home visits, bi-weekly emails, and mailed behaviour supports (intervention group), or 2) Monthly emails with general health information (control group). Primary and secondary outcomes will be assessed at baseline, post-intervention (6-months), and 18-month follow-up, and data will be analyzed by intention to treat.

This study tests a novel and promising approach to obesity prevention - an approach that engages families at home, where they eat, play, and sleep. The interdisciplinary investigator team has partnered with parents and key knowledge users in public health and primary care to develop this intervention. As a result, this research could provide a sustainable model for early life obesity prevention, leading to long-term improvements in health and reduction in costs to the health system and society as a whole.

ELIGIBILITY:
Inclusion Criteria:

* families who have at least 1 child age 18 months - 5 years
* families who live in the Guelph area
* families who can respond to English surveys

Exclusion Criteria:

* plan to move away within the next year
* have children with severe health conditions (e.g., cerebral palsy) that prevent participation in study activities.

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Child - change in BMI | Baseline, 6 Months and 18 Months
  Trained staff will use standard practices to measure child height to the nearest 0.1 cm with a Shorrboard stadiometer and child weight to the nearest 0.1 kg using a Seca scale. BMI will be the ratio of weight (kg) to the square of standing height (m).

SECONDARY OUTCOMES:
Child - change in waist circumference | Baseline, 6 Months, 18 Months
  Trained staff will measure waist circumference at the top of the iliac crest to the nearest 0.1cm, using the NIH protocol.
Child - change in % body fat | Baseline, 6 Months, 18 Months
  Trained staff will use bioelectrical impedance analysis to assess child body composition and use the equation by Kusher to determine % body fat.
Child - change in sleep duration | Baseline, 6 Months, 18 Months
  Sleep duration will be assessed using the wActiSleep+ Activity Monitor (ActiGraph). Activity monitors will be worn on the child's non-dominant wrist for 7 consecutive days. Sleep measures will be determined using the validated Sadeh algorithm.
Child - change physical activity | Baseline, 6 Months, 18 Months
  Physical activity will be assessed using the wActiSleep+ Activity Monitor (Actigraph). Activity monitors will be worn on the child's hip for 7 consecutive days. Validated cut-off values for physical activity for preschool children will be used to determine physical activity.
Child - change in sedentary behaviour | Baseline, 6 Months, 18 Months
  Sedentary behaviour will be assessed using the wActiSleep+ Activity Monitor (Actigraph). Activity monitors will be worn on the child's hip for 7 consecutive days. Validated cut-off values for sedentary behaviour for preschool children will be used to assess sedentary behaviour.
Child - change in dietary behaviour (sugar sweetened beverages, fruit and vegetable intake, etc). | Baseline, 6 Months, 18 Months
  To assess children's dietary intake, parents will be asked record all food and beverages that their child consumes over a 3-days period (2 weekdays and 1 weekend day). Data will be analyzed for energy and nutrient intake via ESHA nutrient analysis software.
Adult and child - change in family meals | Baseline, 6 Months, 18 Months
  Parents will report frequency of family meals using an item from The Home Environment Inventory.
Adult - change in BMI | Baseline, 6 Months, 18 Months
  Trained staff will use standard practices to measure adult height to the nearest 0.1 cm with a stadiometer and adult weight to the nearest 0.1 kg using a Seca scale. BMI will be the ratio of weight (kg) to the square of standing height (m).
Adult - change in waist circumference | Baseline, 6 Months, 18 Months
  Trained staff will measure waist circumference at the top of the iliac crest to the nearest 0.1cm, using the NIH protocol.
Adult - change in % body fat | Baseline, 6 Months, 18 Months
  Trained staff will measure parental body composition using air displacement plethysmography, i.e., BODPOD™.
Adult - change in sleep duration | Baseline, 6 Months, 18 Months
  Sleep duration will be assessed using the wActiSleep+ Activity Monitor (ActiGraph). Activity monitors will be worn on the participants non-dominant wrist for 7 consecutive days. Sleep measures will be determined using the a validated Sadeh algorithm.
Adult - change in physical activity | Baseline, 6 Months, 18 Months
  Physical activity will be assessed using the wActiSleep+ Activity Monitor (Actigraph). Activity monitors will be worn on the participant's hip for 7 consecutive days. Validated cut-off values for physical activity will be used to determine physical activity.
Adult - change in sedentary behaviour | Baseline, 6 Months, 18 Months
  Sedentary behaviour will be assessed using the wActiSleep+ Activity Monitor (Actigraph). Activity monitors will be worn on the child's hip for 7 consecutive days. Validated cut-off values for sedentary behaviour will be used to assess sedentary behaviour.
Adult - change in dietary behaviour | Baseline, 6 Months, 18 Months
  To assess parent's dietary intake, parents will complete one 24-hour recall using the Automated Self-Administered 24-hour-Canada (ASA24®) dietary recall system, a web-based tool that collects and codes 24-hour recalls using the Canadian Nutrient File.
Adult - motivation for lifestyle change | Baseline, 6 Months, 18 Months
  Treatment Self-Regulation Questionnaire will be used to assess family level of autonomous motivation.
Social determinants of obesity | Baseline, 6 Months, 18 Months
  The investigators will assess parental education, marital status, annual household income, parental work patterns, food security, parent perception of neighbourhood safety, and access to grocery stores and indoor and outdoor spaces to be physically active.
Cost-effectiveness of Intervention | Baseline, 6 Months, 18 Months
  The cost effectiveness of the study intervention will be assessed from a societal perspective. The direct costs associated with the intervention will be assessed, as well as health services use and indirect patient costs for both intervention and control groups. Direct costs of the intervention will be estimated from process data collected during the intervention. Through surveys at post-intervention, data will also be collected on costs to families for participating in the intervention, including time spent on home visits and other time costs associated with implementing the intervention recommendations. Health services use will be collected from parents and from linkage with administrative datasets (Ontario Health Insurance Plan). Parents will also be asked to report indirect patient costs, including number of missed school/work days.

CONTACTS AND LOCATIONS:
Overall Officials: Jess Haines, PhD, Principal Investigator — Unviersity of Guelph; David Ma, PhD, Study Director — University of Guelph
Locations (1):
- Univeristy of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacob R, Buchholz AC, Darlington G, Duncan AM, Vallis LA, Chaput JP, Annis A, Nixon M, Irwin JD, Morrow D, Ma DWL, Haines J. Impact of a Home-Based Obesity Prevention Intervention on Children's and Parents' BMI: Findings From the Guelph Family Health Study Randomised Controlled Trial. Pediatr Obes. 2026 Jan;21(1):e70062. doi: 10.1111/ijpo.70062. Epub 2025 Oct 22. PMID 41125536
- [Derived] Ribey SCS, Coyle-Asbil HJ, Osojnicki K, Coyle-Asbil B, Vallis LA, Darlington G, Duncan AM, Ma DWL, Haines J, Buchholz AC. Associations between objectively measured nighttime sleep duration, sleep timing, and sleep quality and body composition in toddlers in the Guelph Family Health Study. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-7. doi: 10.1139/apnm-2024-0244. Epub 2024 Nov 20. PMID 39566036
- [Derived] Yu J, Mahajan A, Darlington G, Buchholz AC, Duncan AM, Haines J, Ma DWL; Guelph Family Health Study. Free sugar intake from snacks and beverages in Canadian preschool- and toddler-aged children: a cross-sectional study. BMC Nutr. 2023 Mar 8;9(1):44. doi: 10.1186/s40795-023-00702-3. PMID 36890595